CLINICAL TRIAL: NCT05704959
Title: Does Povidone-Iodine on Nail Affect Pulse Oximeter Reading?
Acronym: PI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Aynur KOYUNCU, Principal Investigator, Assist Prof, Hasan Kalyoncu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PI
Record Dates: First submitted 2023-01-11; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: HEALTHY INDIVIDUALS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measurement (Other)
  Interventions: Diagnostic Test: povidone iodine

INTERVENTIONS:
Diagnostic Test: povidone iodine — Reference measurements were made simultaneously with two separate calibrated pulse oximeter devices from the index, middle and ring fingers of both hands of the participants. One layer of 10% povidone iodine was applied to the index finger, two layers to the middle finger, and three layers to the ring finger of one hand of the participant's choice. Two pulse oximetry measurements were made with the fingers of the other hand, immediately after the application of povidone-iodine and three minutes later, and it was noted on the data collection form.

SUMMARY:
Povidone iodine is still a commonly used antiseptic in hospitals. Although pulse oximetry measurement is used as an important indicator in hospitals, no study has been found examining the effect of povidone iodine on the nail bed on the pulse oximetry result.

DETAILED DESCRIPTION:
Povidone iodine is still a commonly used antiseptic in hospitals. Although pulse oximetry measurement is used as an important indicator in hospitals, no study has been found examining the effect of povidone iodine on the nail bed on the pulse oximetry result. The aim of this study is to determine the effect of 10% povidone iodine on the nail bed on the oxygen saturation reading in pulse oximetry.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer person
* Healthy person

Exclusion Criteria:

* Patients in hospital
* People with finger loss

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
The effect of 10% povidone iodine in the nail bed on the SpO2 reading of the pulse oximeter | during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided